CLINICAL TRIAL: NCT03165110
Title: US ONYX 2.0 Study: A Clinical Study of the Onyx 2.0 System for Blood Glucose Monitoring in Patients With Diabetes
Brief Title: Evaluation of an Ascensia Diabetes Care Blood Glucose Meter and App System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-PRO-2016-001-01
Record Dates: First submitted 2017-04-07; First posted 2017-05-24 (Actual); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Users of the Onyx Blood Glucose Meter/ app System at home (Experimental): Participants have a diagnosis of either type 1 or type 2 diabetes for at least 6 months and use insulin.
  Interventions: Device: Onyx BG Meter / App System

INTERVENTIONS:
Device: Onyx BG Meter / App System — Subjects with diabetes used the Onyx BG Meter / App System at home and assessed the features of the App.

SUMMARY:
The purpose of this study is to assess the utility of the Contour Diabetes App 2.0 when used with the Contour Next One meter (the Onyx system).

DETAILED DESCRIPTION:
The purpose of this study is to assess the utility of the Contour Diabetes App 2.0 when used with the Contour Next One meter (the Onyx system) in the hands of subjects with type 1 diabetes or insulin-using subjects with type 2 diabetes. It is designed to determine the subjects' self-reported success in utilizing the features of the system. Each feature will be evaluated independently, by including a series of statements about each feature set for which a numerical score or rating will be provided by subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18-75 years, male or female
* Read and understand English
* Have diagnosis of type 1 (goal is 40% to 70%) or insulin-using type 2 diabetes for at least 6 months
* Be taking multiple daily insulin injections (MDI) of at least two pre-meal bolus insulin injections daily or using an insulin pump (Goal is not more than 30% of subjects using insulin pump therapy)
* Performing self-monitoring of blood glucose at home at least twice daily
* Have an iOS mobile device or Android mobile device with Bluetooth capability iOS device: iPod, iPad, or iPhone 5 or later version with iOS 9.x or 10.x software Android: smart phone, software version 6.x. Bluetooth: software version 4.0 or higher
* Agree NOT to update the software on their mobile device until after the study is concluded, as follows:
* No updates of Android device to upcoming Android version 7 (Nougat)
* Be willing to utilize the Contour Next One meter and the Contour Diabetes App 2.0 on personal mobile device which communicates to meter to manage diabetes and be willing to keep a study diary

Exclusion Criteria:

* Known Hemophilia or any other bleeding disorder
* Pregnancy (reported by subject; no pregnancy test required)
* Current user of Contour Next One BGMS including Contour Diabetes App.
* Physical, visual or neurological impairments that would make the person unable to perform testing with the Contour Next One BGMS or to use the Contour Diabetes App
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.

  * Immediate family members are the subject's parents, spouse, children, and siblings, including the parent's spouse; step children and adopted children and their spouses.
  * A competitive medical device company is a company that provides a medical device or components of a device that is related to diabetes. For example, people who are not eligible are those who work for companies that create or manufacture the following (or a company that is in a partnership with a company that provides such devices): lancing devices, blood glucose monitoring systems, continuous glucose monitoring systems, insulin pens, or systems related to the measurement of HbA1c. People who are eligible are those who work for companies associated with products such as wound dressings, medications or dietary products.
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee on the subject disposition form).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 March 2017 - 05 May 2017 AMCR Institute, Escondido CA
Groups:
- Users of the Onyx Blood Glucose Meter/ App System at Home: All participants in the study have a diagnosis of either type 1 or type 2 diabetes for at least 6 months and use insulin in their diabetes management.
  Onyx BG Meter / App System: Subjects with diabetes used the Onyx BG Meter / App System at home and assessed the features of the App.
Period: Overall Study
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Started | 47
Completed | 46
Not Completed | 1
Not completed — Anroid phone software incompatibility | 1

BASELINE CHARACTERISTICS:
Population: 46 people with insulin-dependent diabetes
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
Age, Continuous [Mean (Full Range); unit: years] | 50 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 46
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: Percent of Responses From Persons With Diabetes That 'Strongly Agree' or 'Agree' or 'Neither Agree Nor Disagree' With Questionnaire Statements Regarding Success With Syncing the Reading on the Onyx Glucose Meter and App.
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on the success of syncing the blood glucose value on the meter with the App for the Onyx Glucose Meter and App System. Subjects could respond '1Strongly Agree' or '2Agree' or '3Neither Agree nor Disagree' or '4Disagree' or '5Strongly Disagree' or '6No Opinion'.
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes
Measure: Number; unit: percentage of participants
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
percentage of participants | 89.13

2. Primary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or 'Neither Agree Nor Disagree' With Questionnaire Statements Regarding Success in Accessing and Using Smart Reminders Feature in the Onyx App System
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on accessing and using the Smart Reminders feature in the Onyx App System. Subjects could respond '1Strongly Agree' or '2Agree' or '3Neither Agree nor Disagree' or '4Disagree' or '5Strongly Disagree' or '6No Opinion'.Recognize and use "Smart Reminders"
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes
Measure: Count of Participants; unit: Participants
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
Participants
  Strongly Agree, Agree, or Neither Agree/Disagree | 26
  No opinion | 20

3. Primary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neither Agree Nor Disagree' With Questionnaire Statements Regarding Success at Accessing the Expanded Graph and My Readings View in the Onyx App System
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on the subjects ability to access the Expanded Graph and My Readings views in Onyx App System. Subjects could respond '1Strongly Agree' or '2Agree' or '3Neither Agree nor Disagree' or '4Disagree' or '5Strongly Disagree' or '6No Opinion'.
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes
Measure: Count of Participants; unit: Participants
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
Participants | 46

4. Primary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neither Agree Nor Disagree' With Questionnaire Statements Regarding Success in Interpreting the Expanded Graph and My Readings View in the Onyx App System
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on the subjects ability to interpret the Expanded Graph and My Readings views in Onyx the App System. Subjects could respond '1Strongly Agree' or '2Agree' or '3Neither Agree nor Disagree' or '4Disagree' or '5Strongly Disagree' or '6No Opinion'.
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes
Measure: Count of Participants; unit: Participants
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
Participants | 45

5. Secondary Outcome: Change in HbA1c% From Study Start to End of Study
Description: Laboratory reports were used to compare HbA1c results from subjects at visit 1 with HbA1c results at Visit 2 (end of study). The average change of HbA1c for all subjects at Visit 1 were compared to the average change of HbA1c for all subjects at Visit 2. Lower scores are better outcomes.
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes (1 subject was not included in this analysis due to dropping out of study before Visit 2)
Measure: Least Squares Mean (Full Range); unit: change in HbA1c%
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 45
change in HbA1c%
  Site Visit 1 | 7.7273003 [5.6 to 11]
  Site Visit 2 | 7.6993933 [5.6 to 11]

6. Secondary Outcome: Change in Fructosamine (µmol/L) From Study Start to End of Study
Description: Laboratory reports were used to compare fructosamine results from subjects at visit 1 with frustosamine results at Visit 2 (end of study).
Time Frame: 6 Weeks
Population: 46 people with insulin-dependent diabetes
Measure: Least Squares Mean (Full Range); unit: µmol/L
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
µmol/L
  Visit 1 | 332.8 [211 to 555]
  Visit 2 | 322.7 [211 to 555]

7. Secondary Outcome: Average Change in Subject Body Weight From Study Start to End of Study
Description: The average change in subject body weight from study start (Visit 1) to end of study (Visit 2).
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes
Measure: Least Squares Mean (Standard Deviation); unit: lbs
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
lbs
  Site Visit 1 | 194.4 (59.51)
  Site Visit 2 | 193.8 (59.30)

8. Secondary Outcome: Average Change in Subject BMI From Study Start to End of Study
Description: Subject BMI results at visit 1 were compared with BMI results at Visit 2 (end of study).
Time Frame: 6 weeks
Population: 46 people with insulin-dependent diabetes
Measure: Least Squares Mean (Standard Error); unit: Kg/m^2
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
Kg/m^2
  Site Visit 1 | 29.723913 (0.10903799)
  Site Visit 2 | 29.636304 (0.10903799)

9. Secondary Outcome: Average Change in Total Daily Insulin Dose From Study Start to End of Study
Description: A Subjects' self-reported Total Daily Insulin Doses at visit 1 were compared with their self-reported Total Daily Insulin Doses at Visit 2 (end of study).
Time Frame: 6 weeks
Population: change in insulin dose from visit 1 to visit 2.
Measure: Least Squares Mean (Standard Error); unit: IU
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
Number analyzed (Participants) | 46
IU
  Site Visit 1 | 76.869565 (1.4668160)
  Site Visit 2 | 78.326087 (1.4668160)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Users of the Onyx Blood Glucose Meter/ App System at Home
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 2/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Users of the Onyx Blood Glucose Meter/ App System at Home (N=46)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder Infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT03165110/Prot_SAP_000.pdf